CLINICAL TRIAL: NCT04382599
Title: Designing Impactful Warnings for Sugary Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-0277a
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Added sugar warning message (Experimental): Message displayed on warning labels is: "WARNING: High in added sugar."
  Interventions: Behavioral: Text warning with square background; Behavioral: Text warning with octagon background; Behavioral: Icon warning; Behavioral: Graphic warning
- Weight gain warning message (Experimental): Message displayed on warning labels is: "WARNING: Excess consumption of drinks with added sugar contributes to weight gain."
  Interventions: Behavioral: Text warning with square background; Behavioral: Text warning with octagon background; Behavioral: Icon warning; Behavioral: Graphic warning
- Type 2 diabetes warning message (Experimental): Message displayed on warning labels is: "WARNING: Excess consumption of drinks with added sugar contributes to type 2 diabetes."
  Interventions: Behavioral: Text warning with square background; Behavioral: Text warning with octagon background; Behavioral: Icon warning; Behavioral: Graphic warning
- Heart damage warning message (Experimental): Message displayed on warning labels is: "WARNING: Excess consumption of drinks with added sugar contributes to heart damage."
  Interventions: Behavioral: Text warning with square background; Behavioral: Text warning with octagon background; Behavioral: Icon warning; Behavioral: Graphic warning
- Neutral message (Active Comparator): Message displayed on control label is: "Please refrain from littering."
  Interventions: Behavioral: Text warning with square background; Behavioral: Icon warning; Behavioral: Graphic warning

INTERVENTIONS:
Behavioral: Text warning with square background — The warning message is in white text on a black square background
Behavioral: Text warning with octagon background — The warning message is in white text on a black octagon background
  Arms: Added sugar warning message; Heart damage warning message; Type 2 diabetes warning message; Weight gain warning message
Behavioral: Icon warning — The warning message in in white text on a black background, below an icon that conveys the topic the warning is about
Behavioral: Graphic warning — The warning message in in white text on a black background, below a graphic that conveys the topic the warning is about

SUMMARY:
The goal of this online RCT study is to examine how sugar-sweetened beverage (SSB) health warnings influence US adults' perceptions and reactions. The investigators have the following predictions:

1. SSB warnings will be perceived as more effective than the control (message topic)
2. Icon and graphic warnings will be perceived as more effective than text-only warnings (message type)

The investigators will also examine the interaction of warning topic and warning type, but have no specific hypothesis about this interaction.

Finally, the investigators will test the following predictions about the secondary outcomes:

SSB warnings (vs. control), as well as icon and graphic warnings (vs text.warnings), will lead to lower perceived product healthfulness, lower purchase intentions, and higher cognitive elaboration.

DETAILED DESCRIPTION:
Childhood obesity is a major public health problem in the US among racial and ethnic minorities, including among the US's growing Latino population. One promising but understudied policy for addressing childhood obesity is requiring warnings on the front of sugar-sweetened beverage containers. However, the topic and design of warnings that are most effective in communicating the harms of sugar-sweetened beverages remains unknown. This study assess which warning topics and which warning designs lead to the greatest perceived message effectiveness among US Latino and non-Latino parents of children ages 2-12. The investigators focus on parents as they are the primary decision-makers and purchasers of food products for children and exert strong influence over their children's dietary intake and food attitudes.

Setting: The trial will take place online on a survey developed using Qualtrics.

Recruitment: Participants will be recruited online by CloudResearch PrimePanels, a survey research platform with access to over 20 million participants. As such, participants will have to be PrimePanels members in order to participate.

Informed Consent: After determining eligibility, eligible participants will be directed to a page on Qualtrics with the consent form. Participants acknowledge their consent in the study by clicking the "next page" arrow and proceeding to the study.

Randomization: After consenting, the participant is randomly assigned to to view one of the 5 warning topics. "WARNING: High in added sugar" (added sugar), "WARNING: Excess consumption of drinks with added sugar contributes to weight gain" (weight gain), "WARNING: Excess consumption of drinks with added sugar contributes to type 2 diabetes" (Type 2 diabetes), "WARNING: Excess consumption of drinks with added sugar contributes to heart damage" (heart damage), and "Please refrain from littering" (control). Within each of the four experimental arms, participants see the message displayed on four different types of warning designs: a text warning on a square background, a text warning on a octagon background, and icon warning, and a graphic warning. Within the control arm, participants see the message displayed on three different types of warning designs: a text warning on a square background, an icon warning, and a graphic warning. Participants randomly see the different warning designs in a random order.

Survey: The participants complete a survey answering behavioral perceptions and intentions questions about the different warning labels.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Prime Panels member
* have at least one child ages 2-12
* Currently reside in the US

Exclusion Criteria:

* less than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1078 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Perceived message effectiveness | During survey, which lasts approximately 12-15 minutes.
  Perceived message effectiveness as measured by average response to three statements:
  This message makes me concerned about the health effects of drinking beverages with added sugar. Response options are on a scale (1=Strongly disagree...5=Strongly agree).
  This message makes drinking beverages with added sugar seem unpleasant to me. Response options are on a scale (1=Strongly disagree...5=Strongly agree).
  This message discourages me from wanting to drink beverages with added sugar. Response options are on a scale (1=Strongly disagree...5=Strongly agree).

SECONDARY OUTCOMES:
Perceived product healthfulness of beverages with added sugar | During survey, which lasts approximately 12-15 minutes.
  Measured with the question, "How healthy or unhealthy would it be for your child to drink beverages with added sugar every day?" Response options are on a scale (1= Very unhealthy...5=Very healthy).
Intentions to purchase beverages with added sugar | During survey, which lasts approximately 12-15 minutes.
  Measured with the question, "How likely are you to buy beverages with added sugar for your child in the next four weeks?" Response options are on a scale (1 = Not at all likely...5 = Extremely likely).
Thinking about the health problems from beverages with added sugar | During survey, which lasts approximately 12-15 minutes.
  Measured with the question, "How much does this message make you think about the health problems caused by drinking beverages with added sugar?" Response options are on a scale (1=Not at all...5=Very much).

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Hall, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall MG, Lazard AJ, Grummon AH, Higgins ICA, Bercholz M, Richter APC, Taillie LS. Designing warnings for sugary drinks: A randomized experiment with Latino parents and non-Latino parents. Prev Med. 2021 Jul;148:106562. doi: 10.1016/j.ypmed.2021.106562. Epub 2021 Apr 18. PMID 33878350